CLINICAL TRIAL: NCT00914628
Title: TK008: Randomized Phase III Trial of Haploidentical HCT With or Without an Add Back Strategy of HSV-Tk Donor Lymphocytes in Patients With High Risk Acute Leukemia
Brief Title: Efficacy Study on the Strategy of HSV-Tk Engineering Donor Lymphocytes to Treat Patients With High Risk Acute Leukemia
Acronym: TK008
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: EMA withdrew the marketing Authorisation at the request of AGC Biologics S.p.A (formerly MolMed S.p.A), which decided to permanently discontinue the marketing of the product for commercial reasons
Sponsor: AGC Biologics S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TK008; 2009-012973-37 (Registry Identifier: EUdraCT number)
Record Dates: First submitted 2009-06-03; First posted 2009-06-05 (Estimated); Results first posted 2021-06-22 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Acute Leukemia (Category)
Keywords: high risk acute leukemia; HSV-TK; Haploidentical HCT; GvHD; GvL; Immunoreconstitution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): HSV-TK engineering donor Lymphocytes
  Interventions: Genetic: HSV-Tk
- B (Active Comparator): T-cell depleted or T-cell replete strategies
  Interventions: Other: T-cell depleted or T-cell replete strategies

INTERVENTIONS:
Genetic: HSV-Tk — Infusion of approximately 1±0.2 x 10^7 HSV-Tk genetically modified CD3+ cells/Kg between day +21 and day +49 after haploidentical HCT; in absence of immune reconstitution and GvHD further infusions up to 4 will be administered on monthly basis.
  Arms: A
Other: T-cell depleted or T-cell replete strategies — Haploidentical HCT with the infusion of CD34+ cells plus a fixed dose of T cells (1 x 10^4/Kg) or unmanipulated haploidentical stem cell transplantation followed by high-dose cyclophosphamide as part of GvHD prophylaxis
  Arms: B

SUMMARY:
The main objective of this randomized trial is to compare disease-free survival (DFS) in high risk leukemia patients who underwent haploidentical HCT followed by an add back strategy of HSV-Tk donor lymphocytes or standard haploidentical HCT

DETAILED DESCRIPTION:
Delayed immune-reconstitution remains one of the main limitation of haploidentical stem cell transplantation. The risk of severe infections remains high for several months and CD3+ reconstitution could take more than 10 months. The low number of lymphocytes infused with the graft, the degree of HLA (Human Leukocyte Antigen) disparity, and a reduced thymic function in adults and differences in host/donor antigen presenting cells are contributing causes.

The infusions of HSV-TK engineered lymphocytes may represent a significant therapeutic improvement in haploidentical HCT (hematopoietic cell transplantation), because it remarkably may enhance both GvL (Graft versus Leukemia) activity, thus reducing the occurrence of disease relapse, and post-transplant immune reconstitution in the absence of chronic immune suppression, thus decreasing the rate of both post-transplant opportunistic infections and transplant-related mortality. Furthermore, the efficient control of GvHD achieved via the suicide mechanism allows also the multiple infusion of HSV-TK-treated donor lymphocytes, when needed, that might further improve post-transplant host immune reconstitution, and survival in patients receiving haplo-HCT. Finally, this therapeutic approach can become a valuable option for all candidates, including patients with advanced disease and older age.

The proposed clinical trial represents an innovative therapeutic treatment for patients affected by high risk acute leukemia, who have undergone haploidentical stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Any of the following conditions:

  1. AML and ALL in 1st complete remission (CR1)
  2. AML and ALL in 2nd or subsequent CR
  3. secondary AML in CR
  4. AML and ALL in 1st or 2nd relapse or primary refractory
* Family donor with patient-donor number of HLA mismatches ≥ 2 (full haploidentical), or family donors sharing one HLA-haplotype with the patient
* Stable clinical conditions and life expectancy > 3 months
* PS ECOG < 2
* Serum creatinine < 1.5 x ULN
* Bilirubin < 1.5 x ULN; transaminases < 3 x ULN
* Left ventricular ejection fraction > 45%
* QTc interval < 450 ms
* DLCO > 50%
* Patients, or legal guardians, and donors must sign an informed consent indicating that they are aware this is a research study and have been told of its possible benefits and toxic side effects

Exclusion Criteria:

* Patients with life-threatening condition or complication other than their basic condition
* Contraindication to haploidentical HCT as defined by the Investigator
* Patients with active CNS disease
* Pregnant or lactation.

Exclusion criteria for HSV-Tk infusion:

* Infections requiring administration of ganciclovir or valganciclovir at the time of infusion
* GvHD requiring systemic immunosuppressive therapy
* Ongoing systemic immunosuppressive therapy after haploidentical HCT
* Administration of G-CSF after haploidentical HCT

HSV-Tk cells can be administered after an adequate patient wash-out period (24 hours)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2010-04-12 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Lambiase, MD, Study Director — AGC Biologics S.p.A.
Locations (36):
- United States (3):
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Washington University Medical School, St Louis, Missouri
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
- Belgium (3):
  - Universitair Ziekenhuis, Ghent
  - University Hospitals Leuven, Leuven
  - Centre Hospitalier Universitaire de Liège - Domaine Universitaire du Sart Tilman, Liège
- France (8):
  - Hôpital Jean Minjoz, Besançon
  - Centre Hospitalier Universitaire de Clermont-Ferrand, Clermont-Ferrand
  - Centre Hospitalier Régional Universitaire de Lille, Lille
  - Institut Paoli-Calmettes, Marseille
  - Centre Hospitalier Universitaire de Nantes, Nantes
  - Hôpital l'Archet, Nice
  - Hôpital Saint-Antoine, Paris
  - IUCT Oncopole - Institut Universitaire du Cancer de Toulouse, Toulouse
- Germany (6):
  - Charitè; Campus Benjamin Franklin, Berlin
  - University Medical Center Hamburg-Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - University of Leipzig, Leipzig
  - Universitat Tubingen, Tübingen
  - Medizinische Klinik und Poliklinik, Ulm
- George Papanicolaou Hospital, Thessaloniki, Greece
- Chaim Sheba Medical Center, Tel Litwinsky, Israel
- Italy (9):
  - Azienda Sanitaria Ospedaliera S.Croce e Carle, Cuneo, CN
  - Azienda Ospedaliero-Universitaria Policlinico-Vittorio Emanuele, Catania, CT
  - Azienda Ospedaliera Universitaria Careggi, Florence, FI
  - Azienda Ospedaliera Ospedali Riuniti Villa Sofia - Cervello, Palermo, PA
  - Azienda Ospedaliero-Universitaria Città della Salute e della Scienza di Torino, Presidio Molinette, Torino, TO
  - Ospedale Santa Maria della Misericordia, Udine, UD
  - Policlinico G. B. Rossi, Azienda ospedaliera universitaria integrata di Verona, Verona, VR
  - Ospedale San Raffaele, Milan
  - Azienda Ospedaliero-Universitaria Policlinico di Modena, Modena
- Santaros Klinikos, Vilnius, Lithuania
- Centro Hospitalar Lisboa Norte, E.P.E., Lisbon, Portugal
- Spain (3):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Instituto Catalán de Oncología, L'Hospitalet de Llobregat
  - Hospital de Navarra, Pamplona

IPD SHARING:
Plan to Share IPD: No
No, only information requested by law will be released

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study period:
  Date of First patient enrolled: 12.04.2010; Date of Last patient completed: 30.11.2019; Date of End of study: 30.11.2019.
Pre-assignment Details: Planned sample size n.170; Randomized patients n. 92. Discontinued n. 70; Early termination by the Sponsor n. 22;
Groups:
- A-Experimental Arm: Patients received an infusion of CD34+ cells plus a dose of T cells (approximately 1 x 104/Kg) followed by the infusion of HSV-TK genetically modified CD3+ cells. In absence of immune reconstitution and GvHD further infusions up to 4 will be administered on monthly basis.
  HSV-TK engineering donor Lymphocytes
- B - Control Arm: The physician could choose between the infusion of CD34+ cells plus a dose of T cells (approximately 1 x 104/Kg) or unmanipulated haploidentical transplantation (bone marrow or peripheral blood) followed by high-dose cyclophosphamide.
Period: Overall Study
Arm/Group | A-Experimental Arm | B - Control Arm
Started | 64 (Referred to all randomized patient) | 28 (Referred to all randomized patient)
Completed | 0 (Early termination of the Study) | 0 (Early termination of the Study)
Not Completed | 64 | 28
Not completed — Death | 35 | 17
Not completed — Medical decision | 4 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Lack of Efficacy | 1 | 0
Not completed — non-randomized | 1 | 0
Not completed — Relapse | 1 | 2
Not completed — Study terminated by Sponsor | 14 | 8
Not completed — Patients who did not receive a single dose | 7 | 1

BASELINE CHARACTERISTICS:
Groups:
- A - Experimental Arm: patients received the infusion of CD34+ cells plus a dose of T cells (approximately 1 x 104/Kg), followed by the infusion of HSV-TK genetically modified CD3+ cells In absence of immune reconstitution and GvHD further infusions up to 4 will be administered on monthly basis.
- B- Comparator Arm: the physician chose whether the patient received the infusion of CD34+ cells plus a dose of T cells (approximately 1 x 104/Kg) or an unmanipulated haploidentical bone marrow or peripheral blood transplant followed by high-dose cyclophosphamide.
- Total: Total of all reporting groups
Arm/Group | A - Experimental Arm | B- Comparator Arm | Total
Number analyzed (Participants) | 64 | 28 | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.89 (15.29) | 51.43 (12.41) | 47.58 (14.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 9 | 32
  Male | 41 | 19 | 60
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 0 | 1
  Black | 3 | 1 | 4
  Caucasian | 55 | 24 | 79
  Other | 5 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Disease-free Survival (DFS)
Description: Defined as the measure from the date of randomization until the date of relapse (or progression), or death from any cause, whichever occurs first.
  Disease relapse or progression was determined by the Investigator based on the following disease examination:
  * Morphology (bone marrow or peripheral blood)
  * Confirmation of mixed or full chimerism (evaluation of the degree of chimerism between donor/host, according to institutional clinical practice, on bone marrow or peripheral blood)
  * Cytogenetic and/or molecular and/or other tests, according to institutional clinical practice (bone marrow or peripheral blood).
Time Frame: From the date of randomization, assessed up to 12 months
Population: The analysis has been performed for all patients in the two treatment arms. The NRM analysis was performed on the "Intention to Treat Population" (ITT) and "Per Protocol" (PP) set populations.
Measure: Count of Participants; unit: Participants
Arm/Group | A-Experimental Arm | B - Control Arm
Number analyzed (Participants) | 64 | 28
Participants
  DFS on ITT: Patients with DFS event | 45 | 20
  DFS on ITT: Censored patients | 19 | 8
  DFS on PP Set: number analyzed (Participants) | 38 | 26
  DFS on PP Set: Patients with DFS event | 25 | 18
  DFS on PP Set: Censored patients | 13 | 8
  DFS on ITT - day 21 after transplant: number analyzed (Participants) | 55 | 28
  DFS on ITT - day 21 after transplant: Patients with DFS event | 38 | 20
  DFS on ITT - day 21 after transplant: Censored patients | 17 | 8
  DFS on PP Set day 21 after transplant: number analyzed (Participants) | 38 | 26
  DFS on PP Set day 21 after transplant: Patients with DFS event | 25 | 18
  DFS on PP Set day 21 after transplant: Censored patients | 13 | 8
Statistical Analysis 1: Comparison: A-Experimental Arm vs B - Control Arm; Test type: Superiority; p = 0.8974, Log Rank
Statistical Analysis 2: Comparison: A-Experimental Arm vs B - Control Arm; DFS- Intention-To-Treat population- from baseline to day 21; Test type: Superiority; p = 0.7612, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: A-Experimental Arm vs B - Control Arm; Test type: Superiority; p = 0.5995, Log Rank
Statistical Analysis 4: Comparison: A-Experimental Arm vs B - Control Arm; DFS- Intention-To-Treat population - day 21 after transplant; Test type: Superiority; p = 0.4078, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: A-Experimental Arm vs B - Control Arm; DFS- Per-Protocol Set; Test type: Superiority; p = 0.3351, Log Rank
Statistical Analysis 6: Comparison: A-Experimental Arm vs B - Control Arm; DFS- Per-Protocol Set; Test type: Superiority; p = 0.1233, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: A-Experimental Arm vs B - Control Arm; DFS- Per-Protocol Set DFS-day 21 after transplant; Test type: Equivalence; p = 0.5995, Log Rank
Statistical Analysis 8: Comparison: A-Experimental Arm vs B - Control Arm; DFS- Per-Protocol Set DFS-day 21 after transplant; Test type: Superiority; p = 0.4078, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Overall Survival (OS)
Description: any death without previous occurrence of a documented relapse (or progression).Patients alive or without any follow up will be censored.
Time Frame: From the date of randomization to the date of death, assessed up to 12 months
Population: TThe analysis has been performed for all patients in the two treatment arms. The NRM analysis was performed on the "Intention to Treat Population" (ITT) and "Per Protocol" (PP) set populations.
Measure: Count of Participants; unit: Participants
Arm/Group | A-Experimental Arm | B - Control Arm
Number analyzed (Participants) | 64 | 28
Participants
  OS on ITT: Censored patients | 22 | 10
  OS on ITT: Deaths | 42 | 18
  OS on PP Set: number analyzed (Participants) | 38 | 26
  OS on PP Set: Censored patients | 14 | 10
  OS on PP Set: Deaths | 24 | 16
  OS on ITT- day 21 after transplant: number analyzed (Participants) | 55 | 28
  OS on ITT- day 21 after transplant: Censored patients | 20 | 10
  OS on ITT- day 21 after transplant: Deaths | 35 | 18
  OS on PP Set - day 21 after transplant: number analyzed (Participants) | 51 | 28
  OS on PP Set - day 21 after transplant: Censored patients | 18 | 10
  OS on PP Set - day 21 after transplant: Deaths | 33 | 18
Statistical Analysis 1: Comparison: A-Experimental Arm vs B - Control Arm; Test type: Superiority; p = 0.7660, Log Rank; Statistical analysis was performed on Intention-To-Treat population
Statistical Analysis 2: Comparison: A-Experimental Arm vs B - Control Arm; Statistical analysis has been performed for Intention-To-Treat population; Test type: Superiority; p = 0.6706, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: A-Experimental Arm vs B - Control Arm; Statistical analysis has been performed for Per-Protocol Set); Test type: Superiority; p = 0.7332, Log Rank
Statistical Analysis 4: Comparison: A-Experimental Arm vs B - Control Arm; Statistical analysis has been performed for Per-Protocol Set); Test type: Superiority; p = 0.6439, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Immune Reconstitution (IR)
Description: Assess how many patients experience IR. For the assessment, competing risk analysis was performed considering death, relapse, and disease progression as competing events. Patients who were still alive and had no recovery (IR) nor relapse (or progression) were censored.IR is defined as achieving a level of circulating CD3+ ≥ 100/μL for two consecutive observations. The following laboratory examinations are performed:
  * Hematology: WBC (full and differential), RBC, platelets, Hb, Htc, MCV, MPV, serology CMV (PCR and antigenemia).
  * Blood chemistry: AST, ALT, γGT, total bilirubin, LDH.
Time Frame: Weekly up to IR after engraftment of HCT, monthly for 6 months from date of IR and then at month 9 and 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | A-Experimental Arm | B - Control Arm
Number analyzed (Participants) | 58 | 28
Participants
  IR on ITT: Patients with immune reconstitution without previous relapse or progression | 38 | 22
  IR on ITT: Deaths without previous immune reconstitution, relapse or progression | 13 | 5
  IR on ITT: Patients with relapse or progression without previous immune reconstitution | 6 | 1
  IR on ITT: Censored patients | 1 | 0
  IR on PP Set: number analyzed (Participants) | 38 | 26
  IR on PP Set: Patients with immune reconstitution without previous relapse or progression | 29 | 22
  IR on PP Set: Deaths without previous immune reconstitution, relapse or progression | 4 | 3
  IR on PP Set: Patients with relapse or progression without previous immune reconstitution | 5 | 1
  IR on PP Set: Censored patients | 0 | 0
Statistical Analysis 1: Comparison: A-Experimental Arm vs B - Control Arm; This Statistical analysis refers to Immune reconstitution and was performed by Gray's Test for Equality of Cumulative Incidence Functions for intention-To-Treat population; Test type: Superiority; p = 0.1735, Chi-squared
Statistical Analysis 2: Comparison: A-Experimental Arm vs B - Control Arm; This Statistical analysis refers to deaths without previous immune reconstitution, relapse or progression and was performed by Gray's Test for Equality of Cumulative Incidence Functions for intention-To-Treat population; Test type: Superiority; p = 0.5958, Chi-squared
Statistical Analysis 3: Comparison: A-Experimental Arm vs B - Control Arm; This Statistical Analysis refers to patients with relapse or progression without previous immune reconstitution and was performed Gray's Test for Equality of Cumulative Incidence Functions; Test type: Superiority; p = 0.2889, Chi-squared
Statistical Analysis 4: Comparison: A-Experimental Arm vs B - Control Arm; This Statistical analysis refers to Immune reconstitution and was performed by Gray's Test for Equality of Cumulative Incidence Functions for Per-Protocol Set; Test type: Superiority; p = 0.1642, Chi-squared
Statistical Analysis 5: Comparison: A-Experimental Arm vs B - Control Arm; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = 0.8739, Log Rank
Statistical Analysis 6: Comparison: A-Experimental Arm vs B - Control Arm; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p = 0.2304, Chi-squared

4. Secondary Outcome: Engraftment Rate
Description: Defined as the persistent blood cells count above predefined level.
Time Frame: At day 15 after HCT, monthly for 6 months after HCT and then at month 9 and 12
Population: Due to the early termination of the study, the analysis was not performed because data were not collected for this Outcome Measure
Arm/Group | A - Experimental Arm | B- Comparator Arm
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Cumulative Incidence of Grade 2, 3, or 4 Acute GvHD (aGvHD)
Description: Diagnosed and graded according to standard criteria.
  Grade 1:
  Skin: Stage 1-2: Rash on < 25% of skin or Rash on 25-50% of skin Liver: Stage 1-2: Bilirubin 2-3 mg/dl or Bilirubin 3-6 mg/dl Gastrointestinal: Stage 1-2: Diarrhoea > 500 ml/day or persistent nausea or Diarrhoea > 1000ml/day
Time Frame: from the date of HCT until the date of the first occurrence of aGvHD, assessed up to 6 months
Population: as for outcome 4
Arm/Group | A - Experimental Arm | B- Comparator Arm
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Cumulative Incidence of Chronic GvHD (cGvHD)
Description: Diagnosed and graded according to standard NIH consensus criteria
Time Frame: From the date of HCT until the date of the first occurrence of cGvHD, assessed up to 12 months
Population: as for outcome 4
Arm/Group | A - Experimental Arm | B- Comparator Arm
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Duration of GvHD Episodes
Description: Diagnosed and graded according to standard NIH consensus criteria
Time Frame: From the date of start until the date of resolution and duration of immunosuppressive treatments administered for controlling GvHD assessed up to 12 months
Population: Due to the early termination of the study, the analysis was not performed.because data were not collected for this Outcome Measure
Groups:
- B - Comparator Arm: The physician chose whether the patient received the infusion of CD34+ cells plus a dose of T cells (approximately 1 x 104/Kg) or an unmanipulated haploidentical bone marrow or peripheral blood transplant followed by high-dose cyclophosphamide.
Arm/Group | A - Experimental Arm | B - Comparator Arm
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Cumulative Incidence of Relapse (CIR)
Description: Defined on the basis of morphologic evidence of leukaemia in bone marrow or other sites. Gray's test was used to compare the sub-distribution functions of relapse (or progression) events in the two treatment groups. Patients alive without relapse (or regression) will be censored
Time Frame: from the date of randomization to the date of the first occurrence of relapse, assessed up to 12 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | A-Experimental Arm | B - Control Arm
Number analyzed (Participants) | 64 | 28
Participants
  CIR on ITT population - CIR: Patients with relapse or progression | 18 | 11
  CIR on ITT population - CIR: Deaths without previous relapse or progression | 27 | 9
  CIR on ITT population - CIR: Censored patients | 19 | 8
  CIR on PP Set: number analyzed (Participants) | 38 | 26
  CIR on PP Set: Patients with relapse or progression | 11 | 11
  CIR on PP Set: Deaths without previous relapse or progression | 14 | 7
  CIR on PP Set: Censored patients | 13 | 8
Statistical Analysis 1: Comparison: A-Experimental Arm vs B - Control Arm; This Statistical Analysis refers to ITT Patients with relapse or progression and was performed with Gray's Test for Equality of Cumulative Incidence Functions; Test type: Superiority; p = 0.3526, Chi-squared
Statistical Analysis 2: Comparison: A-Experimental Arm vs B - Control Arm; this Gray's Statistical Analysis refers to ITT Deaths patients without previous relapse or progression and was performed with Test for Equality of Cumulative Incidence Functions; Test type: Superiority; p = 0.4035, Chi-squared
Statistical Analysis 3: Comparison: A-Experimental Arm vs B - Control Arm; this Gray's Statistical Analysis refers to PPS patients with relapse or progression and was performed with Test for Equality of Cumulative Incidence Functions; Test type: Superiority; p = 0.2607, Chi-squared
Statistical Analysis 4: Comparison: A-Experimental Arm vs B - Control Arm; this Gray's Statistical Analysis refers to PPS Deaths patients without previous relapse or progression and was performed with Test for Equality of Cumulative Incidence Function; Test type: Superiority; p = 0.5929, Chi-squared

9. Secondary Outcome: Incidence and Duration of Infectious Episodes and Infectious Disease Mortality
Description: Diagnosis, monitoring and treatment of infectious relevant events
Time Frame: From randomization to the date of resolution, assessed up to 12 months
Population: as for outcome 4
Arm/Group | A - Experimental Arm | B- Comparator Arm
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Evaluate the Acute and Long-term Toxicity Related to the HSV-Tk Infusions
Description: Toxicity profile of HSV-Tk infusions
Time Frame: From HSV-Tk infusions to the date of resolution, assessed up to 12 months
Population: as for outcome 4
Arm/Group | A - Experimental Arm | B- Comparator Arm
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Quality of Life (QoL) and Medical Care Utilization (MCU) in Both Arms
Description: Medical resource use data collected will be used in health economic analyses where it may be combined with other data from other sources such as cost data or other clinical parameters.
Time Frame: from randomization up to 12 months
Population: as for outcome 4
Arm/Group | A - Experimental Arm | B- Comparator Arm
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Non-relapse Mortality (NRM)
Description: Defined for all patients as any death without previous occurrence of a documented relapse (or progression). Absence of relapse was determined by the Investigator based on the following disease examination:
  * Morphology (bone marrow or peripheral blood)
  * Confirmation of mixed or full chimerism (evaluation of the degree of chimerism between donor/host, according to institutional clinical practice, on bone marrow or peripheral blood)
  * Cytogenetic and/or molecular and/or other tests, according to institutional clinical practice (bone marrow or peripheral blood).
  Gray's test was used to compare the sub-distribution functions of the death without previous relapse (or progression) and relapse (or progression) events in the two treatment groups.
Time Frame: From the date of randomization to the date of death, assessed up to 12 months.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | A-Experimental Arm | B - Control Arm
Number analyzed (Participants) | 64 | 28
Participants
  NRM on ITT population: Deaths without previous relapse or progression | 27 | 9
  NRM on ITT population: Patients with relapse or progression | 18 | 11
  NRM on ITT population: Censored patients | 19 | 8
  NRM on PP Set: number analyzed (Participants) | 38 | 26
  NRM on PP Set: Deaths without previous relapse or progression | 14 | 7
  NRM on PP Set: Patients with relapse or progression | 11 | 11
  NRM on PP Set: Censored patients | 13 | 8
Statistical Analysis 1: Comparison: A-Experimental Arm vs B - Control Arm; This Statistical Analysis refers to ITT Deaths without previous relapse or progression and was performed with Gray's Test for Equality of Cumulative Incidence Functions; Test type: Superiority; p = 0.4035, Chi-squared
Statistical Analysis 2: Comparison: A-Experimental Arm vs B - Control Arm; This statistical test refers to Patients with relapse or progression and was performed to Gray's Test for Equality of Cumulative Incidence Functions; Test type: Superiority; p = 0.3526, Chi-squared
Statistical Analysis 3: Comparison: A-Experimental Arm vs B - Control Arm; This Statistical Analysis refers to PPS Deaths without previous relapse or progression and was performed with Gray's Test for Equality of Cumulative Incidence Functions; Test type: Superiority; p = 0.5929, Chi-squared
Statistical Analysis 4: Comparison: A-Experimental Arm vs B - Control Arm; [analysis description as in outcome 12, analysis 2]; Test type: Superiority; p = 0.2607, Chi-squared

ADVERSE EVENTS:
Time Frame: From day 21 through day 180 or at least 30 days after last dose of HSV-TK.
Description: Safety analyses, Serious Adverse Events and all cause of mortality evaluations were performed on the STDP. STDP is defined as all randomized patients who received at least one haploidentical HCT (80 total patients).
Groups:
- A-Experimental Arm: Analysis performed only on Standard Population so, all randomized patients who received at least an infusion of CD34+ cells plus a dose of T cells (approximately 1 x 104/Kg) followed by the infusion of HSV-TK genetically modified CD3.
  A total of 53/80 were included in the analysis
- B - Control Arm: Analysis performed only on Standard Population. The physician could choose between the infusion of CD34+ cells plus a dose of T cells (approximately 1 x 104/Kg) or unmanipulated haploidentical transplantation (bone marrow or peripheral blood) followed by high-dose cyclophosphamide.
  A total of 27/80 were included in the analysis
Arm/Group | A-Experimental Arm | B - Control Arm
All-Cause Mortality (participants affected / at risk) | 35/53 | 17/27
Serious Adverse Events (participants affected / at risk) | 35/53 | 17/27
Other Adverse Events (participants affected / at risk) | 22/53 | 0/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | A-Experimental Arm (N=53) | B - Control Arm (N=27)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Moderate Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Life threatening Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Life threatening Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Severe Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 | 0
Severe Thymic cyst (Blood and lymphatic system disorders) | 0 | 1
Mild Abdominal pain (Gastrointestinal disorders) | 1 | 0
Severe Colitis (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Severe Stomatitis (Gastrointestinal disorders) | 0 | 1
Severe Vomiting (Gastrointestinal disorders) | 1 | 1
Moderate Pyrexia (General disorders) | 1 | 0
Severe Pyrexia (General disorders) | 1 | 0
Mild Acute graft versus host disease (Immune system disorders) | 1 | 0
Moderate Acute graft versus host disease (Immune system disorders) | 5 | 3
Severe Acute graft versus host disease (Immune system disorders) | 3 | 1
Mild Chronic graft versus host disease (Immune system disorders) | 0 | 1
Moderate Chronic graft versus host disease (Immune system disorders) | 3 | 0
Severe Chronic graft versus host disease (Immune system disorders) | 3 | 1
Moderate Graft versus host disease (Immune system disorders) | 0 | 1
Severe Graft versus host disease (Immune system disorders) | 1 | 0
Severe Anal abscess (Infections and infestations) | 1 | 0
Severe Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0
Severe Cystitis klebsiella (Infections and infestations) | 1 | 0
Moderate Cystitis viral (Infections and infestations) | 1 | 1
Severe Cytomegalovirus colitis (Infections and infestations) | 1 | 0
Cytomegalovirus colitis Cytomegalovirus colitis (Infections and infestations) | 1 | 0
Severe Cytomegalovirus infection (Infections and infestations) | 1 | 1
Severe Cytomegalovirus viraemia (Infections and infestations) | 1 | 0
Moderate Device related infection (Infections and infestations) | 1 | 0
Severe Device related infection (Infections and infestations) | 0 | 1
Moderate Epstein-Barr virus infection (Infections and infestations) | 1 | 1
Severe Epstein-Barr virus infection (Infections and infestations) | 1 | 0
Moderate Gastroenteritis (Infections and infestations) | 0 | 1
Moderate Herpes zoster infection neurological (Infections and infestations) | 1 | 0
Severe Lung infection pseudomonal (Infections and infestations) | 0 | 1
Moderate Otitis media acute (Infections and infestations) | 1 | 0
Severe Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0
Moderate Pneumonia (Infections and infestations) | 1 | 1
Severe Pneumonia (Infections and infestations) | 3 | 0
Life threatening pneumonia (Infections and infestations) | 0 | 1
Severe Pneumonia cytomegaloviral (Infections and infestations) | 1 | 0
Moderate Pneumonia klebsiella (Infections and infestations) | 1 | 0
Severe Pneumonia klebsiella (Infections and infestations) | 0 | 1
moderate Pneumonia pseudomonal (Infections and infestations) | 0 | 1
Severe Salmonellosis (Infections and infestations) | 1 | 0
Life threatening Sepsis (Infections and infestations) | 0 | 1
Life threatening Septic shock (Infections and infestations) | 0 | 2
Severe Skin infection (Infections and infestations) | 1 | 0
Severe Soft tissue infection (Infections and infestations) | 0 | 1
Moderate Staphylococcal infection (Infections and infestations) | 0 | 1
Severe Systemic candida (Infections and infestations) | 1 | 0
Life threatening Toxoplasmosis (Infections and infestations) | 0 | 1
Severe Transaminases abnormal (Investigations) | 0 | 1
Severe Cachexia (Metabolism and nutrition disorders) | 1 | 0
Life threatening Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Severe Dehydration (Metabolism and nutrition disorders) | 1 | 0
Severe Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Life threatening Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Severe Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Severe Epstein-Barr virus associated lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Severe Leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Life threatening leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Severe Post transplant lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
moderate Dizziness (Nervous system disorders) | 1 | 0
severe Epilepsy (Nervous system disorders) | 0 | 1
moderate Neuropathy peripheral (Nervous system disorders) | 1 | 0
Mild Haematuria (Renal and urinary disorders) | 0 | 1
Life threatening Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Severe Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Severe Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Severe Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Mild Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Life threatening Shock (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | A-Experimental Arm (N=53) | B - Control Arm (N=27)
related to HSV-TK cells (Investigations) | 22 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-23): https://cdn.clinicaltrials.gov/large-docs/28/NCT00914628/Prot_SAP_000.pdf